CLINICAL TRIAL: NCT04843306
Title: "Real-time Augmented Reality Coaching for the Breath-Hold Technique for Pancreatic SBRT Patients"
Brief Title: Breath-Hold Technique for Pancreatic Stereotactic Body Radiation Therapy (SBRT) Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical difficulties that were not able to be resolved.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: J20119; IRB00265565 (Other: JHM IRB)
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: This will be a prospective, randomized, and non-blinded trial to assess the benefit of xR technology for patient education, coaching, and comfort during radiation treatment of pancreatic cancer. Prior to any use of the xR platform for patients, the investigators will perform several dry runs with the Radiation Oncology Physics department to confirm the device and platform can be used safely.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABC technique plus biofeedback (Experimental): Patients will utilize biophysical feedback and coaching during the planning and treatment sessions for radiotherapy to help patients with the ABC technique.
  Interventions: Behavioral: Biofeedback; Behavioral: Active Breathing Control Technique
- Standard of care ABC technique. (Active Comparator): Patients will standard of care instructions for using the ABC technique during the planning and treatment sessions for radiotherapy.
  Interventions: Behavioral: Active Breathing Control Technique

INTERVENTIONS:
Behavioral: Biofeedback — Relaxation coaching will be used in this study.
  Arms: ABC technique plus biofeedback
Behavioral: Active Breathing Control Technique — Active breathing control (ABC) requires patients to reproducibly perform multiple deep-inspiratory breath holds during treatment.

SUMMARY:
The Investigator proposes the development of an extended reality (xR) training platform for patients undergoing radiation treatment for pancreatic cancer. The Investigator wants to investigate the ability of this technology to provide biophysical feedback and coaching during the planning and treatment sessions to help patients with the ABC technique to improve motion management outcomes and reduce treatment related anxiety.

DETAILED DESCRIPTION:
Pancreatic cancer (PCa) is a devastating diagnosis with one of the lowest 5-year overall survival rates of all malignancies. It is estimated that at least 45,000 Americans will die of this disease in 2019, making it the third most common cause of oncologic death. Of the patients that present without evidence of distant spread at the time of diagnosis, only a minority of patients are able to proceed directly to surgical resection which remains the mainstay treatment modality. Historical outcomes show that 30-40% of patients present with borderline resectable (BRPC) or locally advanced (LAPC) disease due to tumor involvement of local vasculature which prevents the patients from proceeding directly to surgery. In this context, neoadjuvant therapy with radiation is often administered in an attempt to downstage tumors prior to surgery, reduce the risk of a margin positive failure, and reduce the risk of local recurrence after surgery. For patients who are truly technically or medically unresectable, radiation can be offered with the intent of providing durable local control. Indeed, a recent autopsy study showed that 30 % of patients who expire from PCa do so due to the locally destructive spread from this disease, highlighting the imperative need for an optimal local control strategy.

Delivering radiation to the pancreas is technically challenging and must be carefully delivered given the risk of injury to radiosensitive organs at risk (OAR) in close proximity such as the bowel and stomach. Compounding this difficulty is the variation in positioning of the tumor and OARs due to respiratory induced motion and variation in bowel gas patterns. To achieve daily accuracy in tumor localization, the investigators employ a comprehensive strategy including strict immobilization, endoscopically placed fiducials, and daily on-board cone beam CT (CBCT). Moreover, the investigators utilize active breathing control (ABC), which requires patients to reproducibly perform multiple deep-inspiratory breath holds during treatment. Radiation to the pancreas is delivered only when the patient is holding patient's breath. During ABC, patients breathe through a snorkel-like device that records the volume of air inhaled during each breath. In this apparatus is a valve that will cut off the flow of air once the inhalation volume passes a certain threshold to ensure the same amount of volume is taken in each time a breath hold is performed. Patients are asked to press on a button to start the recording aspect of the device and then to take a deep breath hold. Once patients reach the desired threshold for the inhaled volume, the valve prevents any further air from being inhaled in, and the patient is asked to hold patient's breath for a duration of 20 - 30 seconds. The treatment team is not present in the room with the patient because of radiation exposure so it requires the patient to follow a series of with the treatment team over an intercom system. Patients are asked to do this without any visual biophysical feedback of patient's waveforms, and to do this repeatedly for multiple times per treatment session. The series of instructions can be challenging for many patients, potentially leading to prolonged treatment times and additional breath holds especially in the early fractions before patients become more familiar with the system. Furthermore, with only one planning session to become acquainted with the ABC device and treatment instructions, patients have limited practical time to gain mastery before returning for patient's actual treatment sessions. This is of concern since patients who struggle with the ABC technique may have less consistent reproducibility of daily tumor positioning which may lead to poorer radiation treatment outcomes.

The Investigator proposes the development of an extended reality (xR) training platform for patients undergoing radiation treatment for pancreatic cancer. The Investigator wants to investigate the ability of this technology to provide biophysical feedback and coaching during the planning and treatment sessions to help patients with the ABC technique to improve motion management outcomes and reduce treatment related anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Patients with a histologically confirmed diagnosis of pancreatic cancer with borderline resectable or locally advanced disease
* Receiving stereotactic body radiation therapy for pancreatic cancer with active breathing control (ABC)
* Able to read and write in English or able to understand/answer study questions and instructions with the aid of an interpreter

Exclusion Criteria:

* Patients who do not provide informed consent
* Patients who chose not to answer the study questions
* Patients who chose not to use the xR device and platform
* Patients with a seizure history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Effectiveness of motion management for SBRT for pancreatic cancer with real-time coaching for the ABC procedure using an augmented reality platform | Up to 3 months from final SBRT session
  The mean range of intra-fraction variation (in millimeters) will be used in assessing the effectiveness of motion management. The result will be compared to historical controls in a "pick the winner" design.

SECONDARY OUTCOMES:
Quality of patient confidence with the ABC procedure with real-time coaching using an augmented reality platform during SBRT for pancreatic cancer as assessed by patient reported outcome measures (PROMs) | Up to 3 months from final SBRT session
  Patient confidence will be assessed with PROMs and the mean score for all patients treated in AR mode 1 will be compared to the mean score for all patients treated in AR mode 2. This PROM consists of 8 questions on a 5-point Likert scale to assess the patient's confidence in performing the ABC procedure with AR mode 1 or 2, and total score ranges from 0 to 32 with higher score signifying greater confidence.
Anxiety of patient with the ABC procedure with real-time coaching using an augmented reality platform during SBRT for pancreatic cancer as assessed by patient reported outcome measures (PROMs) | Up to 3 months from final SBRT session
  Patient anxiety will be assessed with PROMs and the mean score for all patients treated in AR mode 1 will be compared to the mean score for all patients treated in AR mode 2. This PROM consists of 20 questions on a 4-point Likert scale to assess patient anxiety with the ABC procedure and total score ranges from 20 to 80 with higher scores signifying greater anxiety with the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Amol Narang, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States